CLINICAL TRIAL: NCT00648544
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fed, Bioequivalence Study of Pravastatin Sodium 80 mg Tablets Versus Pravachol® 80 mg Tablets In Normal Healthy Non-Smoking Male and Female Subjects
Brief Title: Fed, Bioequivalence Study of Pravastatin Sodium 80 mg Tablets Versus Pravachol® 80 mg Tablets In Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Genpharm ULC (Industry)
Responsible Party: Elliot Offman, Director, Biopharmaceutics, Genpharm ULC
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2722
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pravastatin
- 2 (Active Comparator)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Single-dose 80 mg oral immediate-release tablet
  Arms: 1
Drug: Pravastatin — Single-dose 80 mg oral immediate-release tablets
  Other Names: Pravachol®
  Arms: 2

SUMMARY:
This study was designed to compare the rate and extent of absorption of pravastatin sodium from the following formulations under fed conditions:

1. Pravastatin Sodium 80 mg Tablets (Genpharm Inc. Canada)
2. Pravachol® 80 mg Tablets (Bristol-Myers Squibb Co., U.S.A.) Bioequivalence of these formulations was assessed for pravastatin.

Based on the results from this study, these two 80 mg pravastatin tablet formulations demonstrated bioequivalence under the single-dose fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the following criteria may be included in the study:
* Non-smoking male or female with a minimum age of 18 years.
* Body Mass Index (BMI = weight/height2) greater than or equal to 19 kg/m2 and less than or equal to 26 kg/m2.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.
* Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats/min and temperature between 35.8°C and 37.5°C).
* Negative for drugs of abuse, nicotine , alcohol, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum ß-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides they are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded:
* Known history of hypersensitivity to pravastatin sodium (e.g. Pravachol®, Lipostat®) and/or related drugs such as simvastatin (Zocor®), atorvastatin (Lipitor™), cerivastatin (Baycol®) or fluvastatin (Lescol®).
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the Principal Investigator, or medical designate.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of any significant physical or organ abnormality.
* Any subject with a history of drug abuse.
* Any psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of over-the-counter (OTC) medication within seven days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of oral contraceptives or contraceptive implants (such as Norplant®) within 30 days prior to drug administration or a depot injection of progestogen drug (e.g. Depo-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Any subject who has had blood withdrawals within 56 days preceding this study, taken during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Significant or recent history of asthma (after 12 years of age).
* Any subject with a recent (less than one year) history of alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-07; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic Bioequivalence | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tam, MD, Principal Investigator — Biovail Contract Research
Locations (1):
- Biovail Contract Reseach, Toronto, Ontario, Canada

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html